CLINICAL TRIAL: NCT06036745
Title: An Exploratory Single-Arm, Single-Center Study of Pembrolizumab in Combination With SOX Regimen for Adjuvant Treatment of Stage IIIB-IIIC Gastric Cancer
Brief Title: Exploratory Single-arm, Single-center Adjuvant Treatment of Stage IIIB-IIIC Gastric Cancer With Combination of Palizumab and SOX Regimen
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Adjuvant K+SOX
Record Dates: First submitted 2023-09-07; First posted 2023-09-14 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer Stage IIIB-IIIC
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pembrolizumab + SOX (Experimental)
  Interventions: Drug: Pembrolizumab + SOX

INTERVENTIONS:
Drug: Pembrolizumab + SOX — Pembrolizumab 200mg, ivdrip, q3w; Oxaliplatin 135mg/m2, ivdrip，q3w; Trastuzumab 40 mg/m2，po bid，d1~d14，q21d. Each cycle consists of three weeks, totaling eight cycles

SUMMARY:
it is an an Exploratory Single-Arm, Single-Center Study of Pembrolizumab in Combination with SOX Regimen for Adjuvant Treatment of Stage IIIB-IIIC Gastric Cancer

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects voluntarily join the study and sign an informed consent form; 2. Male or female patients between the ages of 18-75; 3. Adenocarcinoma of the gastric/esophagogastric junction after radical resection was staged at stage IIIB-IIIC; 4. The molecular pathology of gastric cancer must meet at least one of the following three conditions:

  1. Consistent with high-frequency microsatellite instability MSI-H
  2. Consistent with high tumor mutation load TMB-H (≥10 mutations/megabases)
  3. High expression of PD-L1 (CPS score ≥5) 5. Expected survival time > 6 months； 6. ECOG (Eastern US Cooperative Oncology Group) score: 0-1 points; 7. Have not received anti-tumor immunotherapy; 8. Agree to provide archived tumor tissue samples for molecular testing; 9. Have good organ function:

  <!-- -->

  1. Hemoglobin ≥90g/L;
  2. Absolute neutrophil count ≥1.5×109/ L;
  3. Platelet count ≥100×109/ L;
  4. aspartate or alanine aminotransferase ≤ 2.5 times the upper limit;
  5. alkaline phosphatase ≤ 2.5 times the upper normal limit ; 10. Women of reproductive age who need to use a medically approved contraceptive method (such as an IUD, contraceptive pill, or condom) during the study treatment period and for 3 months after the end of the study treatment period; For men who agreed to use an appropriate method of contraception during the trial and for 3 months after the last dose of the trial drug.

     11. Women of reproductive age must be negative for serum or urine HCG within 72 hours prior to study entry. And must be non-lactating.

     Exclusion Criteria:

  <!-- -->

  1. Patients with severe hypertension and poor drug control;
  2. Patients with difficulty in taking oral drugs due to dysphagia, complete or incomplete digestive tract obstruction, active gastrointestinal bleeding, perforation, etc.;
  3. People who are known to be allergic to the ingredients in the test drug or have metabolic disorders;
  4. Simultaneously participating in other tumor experimental drugs or being in other tumor clinical trials.
  5. Severe liver disease (such as cirrhosis, etc.), kidney disease, respiratory disease or uncontrollable diabetes, hypertension and other chronic system diseases; Clinically obvious heart disease, such as congestive heart failure, obvious coronary heart disease, medically difficult to control arrhythmia, hypertension, or myocardial infarction within 6 months, or cardiac insufficiency;
  6. Patients with peripheral nervous system disorders or a history of obvious mental disorders and central nervous system disorders;
  7. Diagnosed with immunodeficiency or received systemic hormone therapy or other forms of immunosuppressive therapy within 7 days prior to initial administration;
  8. Active period > CTCAE (Version 5.0) grade 2 clinical severe infection;
  9. Pregnant and lactating women, women of childbearing age and their spouses refuse to take effective contraceptive methods;
  10. Persons without legal capacity, whose medical or ethical reasons affect the continuation of the research.
  11. Other conditions determined by the investigator to be unsuitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3 years
  the time from the start of surgery to the incurable resection, local recurrence or metastasis, or death from any cause.

SECONDARY OUTCOMES:
Overall survival | 3 years
  the time from the start of surgery to death due to any cause.
perioperative complications | the time from the start of enrollment to 3 months after surgery
  perioperative complications
Adverse Events | the time from the start of enrollment to 90 days after using drugs/ 30 days after surgery
  occurs after a clinical trial subject receives a drug, but is not necessarily causally related to the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China